CLINICAL TRIAL: NCT00586755
Title: Intensive Induction Therapy Followed by Early High Dose Chemotherapy and Bone Marrow Transplantation for Mantle Cell Lymphoma
Brief Title: Intensive Induction Therapy Followed by High Dose Chemo and BM Transplant for Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2165
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Mantle Cell Lymphoma
Keywords: Intensive Induction; High Dose Chemotherapy; Bone Marrow Transplantation; Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intensive Induction-BMT (Experimental): Patients will undergo induction regimen and stem cell mobilization with cyclophosphamide for bone marrow transplant (BMT). This will be immediately followed by high dose therapy with stem cell support.
  Interventions: Procedure: Intensive Induction-BMT

INTERVENTIONS:
Procedure: Intensive Induction-BMT — Patients will undergo an induction regimen consisting of 1 cycle of cytarabine (3 gm/m2 intravenously over 1 hour every 12 hours for 8 total doses) and mitoxantrone (10 mg/m2/d intravenously over 30 minutes daily on days 1, 2, and 3). This will be combined with Alemtuzumab (anti-CD52 antibody) for 6-8 weeks. If, after this one cycle, subjects have not had progression of disease as noted on physical exam or radiographic scans, they will proceed to stem cell mobilization with cyclophosphamide. This will be immediately followed by high dose therapy with stem cell support. Following count recovery, rituximab will be used for 8 total doses as consolidation therapy. Involved field irradiation may be given post-transplant to those with localized bulky disease as well.

SUMMARY:
Patients with mantle cell lymphoma have a grave prognosis. They usually have an initial response to therapy, however progress early in the course of the disease and have very poor survival. We hypothesize that the emergence of drug resistance is responsible for this early failure of therapy and therefore intensive therapy at induction followed by high dose therapy immediately may produce a better outcome.

DETAILED DESCRIPTION:
Subjects will undergo an induction regimen consisting of 1 cycle of cytarabine (3 gm/m2 Intravenously over 1 hour every 12 hours for 8 total doses) and mitoxantrone (10 mg/m2/d intravenously [IV] over 30 minutes daily on days 1, 2, and 3). This will be combined with Alemtuzumab (anti-CD52 antibody) for 6-8 weeks. If, after this one cycle, subjects have not had progression of disease as noted on physical exam or radiographic scans, they will proceed to stem cell mobilization with cyclophosphamide. This will be immediately followed by high dose therapy with stem cell support. Following count recovery, rituximab will be used for 8 total doses as consolidation therapy. Involved field irradiation may be given post-transplant to those with localized bulky disease as well. Day -6: Carmustine (BCNU): 15 mg/kg (or 550 mg/m2) IV over 2 hrs. Day -4: Etoposide Day -2: Cyclophosphamide 100 mg/kg in 1 liter D5W over 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Must have biopsy proven mantle cell lymphoma confirming mantle cell lymphoma. (Flow cytometry, and cyclin D1 or t (11;14) tests of disease site should be done if available at some time in the patient's course before this therapy)
* Radiologic staging studies may be performed up to 6 weeks prior to starting therapy and not be repeated if the treating physician feels it unnecessary
* No other prior malignancy is permitted except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for one year.
* Age > or = to 18 years of age
* For patients who are in first remission from a prior regimen, at least 3 weeks must elapse from a prior chemotherapy and at least 1 week from radiation or antibody therapy.

Exclusion Criteria:

* Significant medical and/or psychiatric illness which, in the opinion of the investigators, may compromise any aspect of the planned treatment.
* The patient cannot have been exposed to chemotherapy to treat any of these diseases (other than mantle cell lymphoma) for at least 3 years prior to entry on this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 1998-02; Primary Completion 2007-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | 1 year
  Number of patients who did not have documented recurrence for at 1 year after bone marrow transplantation.
  We would like to detect an improvement over 0.25 in DFS at one year. Thirty (30) patients will be accrued and complete the transplant phase of therapy. We anticipate only 50% of patients enrolling to complete transplant, noting that approximately 60 patients total will need to be accrued. With 30 patients we can detect an improvement as small as 17% in magnitude, i.e., from an assumed 1-year DFS of 25% to a 1-year DFS of 42% with approximately 80% power. This is based on a one-sided test of hypothesis, testing at significance level 0.05 and the assumption that the true underlying 1-year DFS is 0.25. Greater differences in DFS are expected. If the 1-year DFS with the new treatment is greater than 42% the power is increased.
Progression Free Survival (PFS) | 1 year
  The number of patients who did not have disease progression, recurrence or die for 1 year after bone marrow transplantation.

SECONDARY OUTCOMES:
Response to the induction regimen | 12 weeks
  Number of patients who respond to transplant. Complete Response (CR): No measurable disease. Remission must last for more than 4 weeks.
  Complete Response with Residual Abnormality: CR with persistent mass in the mediastinum or abdomen that has regressed >50% following therapy and then stabilized with NO change over the rest of therapy.
  Partial Response (PR): Reduction of >50% in the sum of the products of the perpendicular diameters of all measurable lesions lasting more than 4 weeks. Disappearance of constitutional symptoms must occur. >30% reduction in extension of the liver below the costal margin at the midclavicular line and the xiphoid process and normalization of liver function tests.
  Stable Disease (SD): < 50% decrease or < 25% increase in the sum of the perpendicular diameters of measurable lesions and no new lesions.
  Progressive Disease (PD): >= 25% increase in the product of the perpendicular diameters of any lesion or new areas of malignant disease.
Response to the transplant phase of therapy | 2 years
  Number of patients who respond to transplant. Complete Response (CR): No measurable disease. Remission must last for more than 4 weeks.
  Complete Response with Residual Abnormality: CR with persistent mass in the mediastinum or abdomen that has regressed >50% following therapy and then stabilized with NO change over the rest of therapy.
  Partial Response (PR): Reduction of >50% in the sum of the products of the perpendicular diameters of all measurable lesions lasting more than 4 weeks. Disappearance of constitutional symptoms must occur. >30% reduction in extension of the liver below the costal margin at the midclavicular line and the xiphoid process and normalization of liver function tests.
  Stable Disease (SD): < 50% decrease or < 25% increase in the sum of the perpendicular diameters of measurable lesions and no new lesions.
  Progressive Disease (PD): >= 25% increase in the product of the perpendicular diameters of any lesion or new areas of malignant disease.
Toxicity of the trial | 2 years
  Number of grade 3 or higher events related to study treatment. Toxicities were assessed using the National Cancer Institute's Common Terminology Criteria for Adverse Events, version 2.0.
Overall Survival (OS) | 5 years
  Number of years patients survived after bone marrow transplantation

CONTACTS AND LOCATIONS:
Overall Officials: David Rizzieri, MD, Principal Investigator — Duke University Health Systems